CLINICAL TRIAL: NCT01889420
Title: Phase I Trial of Everolimus, Pomalidomide and Dexamethasone in Patients With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 1304
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Myeloma in Relapse
Keywords: myeloma; relapse; refractory; relapsed; pomalidomide; pomalyst; everolimus; afinitor; dexamethasone
MeSH Terms: conditions — Neoplasms, Plasma Cell; Recurrence | interventions — Combined Modality Therapy; pomalidomide; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination therapy (Experimental): Pomalidomide: 1 tablet orally, daily for 21 days of a 28 day cycle (dose per cohort) Everolimus: 1 tablet orally for 21 days of a 28 day cycle (dose as per cohort) Dexamethasone 40 mg (20 mg >75yrs) orally, days 1, 8,15, 22 of a 28 day cycle
  Interventions: Drug: Combination therapy

INTERVENTIONS:
Drug: Combination therapy — Following determination of the maximum tolerated dosages in the phase I portion of this study, all patients enrolled in the extension portion will receive the predetermined dosage combination of pomalidomide, everolimus and dexamethasone.
  Cycles will span 28 days. Dosage schedules will be:
  1. Everolimus daily for 28 days of a 28 day cycle;
  2. Pomalidomide daily for 21 days of a 28 day cycle
  3. Dexamethasone once weekly (on days 1,8,15,22) of a 28 day cycle.
  Other Names: Pomalyst; Afinitor

SUMMARY:
This study is being conducted to test the possibility that a combination of three drugs, pomalidomide and everolimus with dexamethasone, may improve patient responses when compared with use of either drug alone, with dexamethasone in refractory/relapsed multiple myeloma.

DETAILED DESCRIPTION:
Given that pomalidomide is an FDA approved drug for patients with relapsed or progressive myeloma, and everolimus has been shown to have single agent activity in relapsed myeloma, it seems reasonable to combine these two active drugs in patients with relapsed/refractory disease. Given that low dose dexamethasone dramatically improved the response rate of pomalidomide, this drug will be added to the combination.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years

Relapsed or progressive multiple myeloma (MM) (Progressive Disease), defined as a 25% increase from the lowest response value in ANY of the following:

Serum M-protein (absolute increase ≥0.5 g/dL)

Urine M-protein (absolute increase of ≥200 mg/24 hours)

Bone marrow plasma cell percentage (≥ 10% absolute increase) in absence of measurable M-protein

Difference in kappa & lambda free light chain levels (ratio must be abnormal; absolute change must be >10 mg/dL)

Patients are also considered to have progressive disease when:

New bone or soft tissue lesions (e.g. plasmacytomas) are identified; or

There is an unequivocal increase in the size of previously existing lesions; or

The development of an otherwise unexplained serum calcium >11.5 mg/dL

Have received 1, but no more than 4 prior treatment regimens or lines of therapy for MM (Induction therapy followed by stem cell transplant & consolidation/maintenance therapy will be considered as one line of therapy)

ECOG Performance status 0 - 2

Life expectancy of at least 12 weeks

Evaluable MM with, at least one of the following, assessed within 21 days prior to randomization:

Serum M-protein ≥ 0.5 g/dL, or Urine M-protein ≥ 200 mg/24 hour, or

In absence of detectable serum or urine M-protein, serum FLC (SFLC) > 100 mg/L (involved light chain) and/or an abnormal kappa/lamda ratio (>4:1 or <2:1), or

Monoclonal plasma cells in a bone marrow biopsy/aspirate of >5%

Adequate organ and marrow function as defined below:

* Leukocytes ≥ 2,500/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin < 2 X ULN
* AST(SGOT)/ALT(SPGT) ≤ 2.5 X ULN
* Creatinine < 1.5 X ULN

Contraception Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for duration of study, and for 90 days after completion of therapy.

A female of child-bearing potential is considered to be any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* No hysterectomy or bilateral oophorectomy; or
* Not naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Male patients must use an effective barrier method of contraception during study and for 3 months following the last dose if sexually active with a female of child-bearing potential.

No prior therapy with pomalidomide or everolimus.

Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.

Receiving any other investigational agents. Minimum 4 week "washout" period is required.

History of allergic reactions attributed to compounds of similar chemical or biologic composition to pomalidomide, everolimus, or other agents used in the study.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Pregnant or nursing (due to the rick for congenital abnormalities and the potential of this regimen to harm nursing infants).

Glucocorticoid therapy (prednisone > 30 mg/day or equivalent) within 14 days prior to randomization.

POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).

Plasma cell leukemia or circulating plasma cells ≥ 2 × 10^9/L.

Waldenstrom's Macroglobulinemia.

Patients with known amyloidosis.

Focal radiation therapy within 7 days prior to randomization. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to randomization (i.e., prior radiation must have been to less than 30% of the bone marrow).

Immunotherapy within 21 days prior to randomization.

Myelodysplastic syndrome

Major surgery (excluding kyphoplasty) within 28 days

Known cirrhosis.

Significant neuropathy (Grades 3 to 4, or Grade 2 with pain) within 14 days

Ongoing graft-vs-host disease.

Using CYP3A4 inhibitors such as Ketoconazole, Ritonavir, Itraconazole, Erythromycin, Clarithromycin, Nelfinavir, Fluconazole, Amiodarone, Cyclosporine, Diltiazem, nefazadone,fluvoxamine, verapamil, chloramphenicol, Indinavir or saquinavir within 7 days of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, MD, Principal Investigator — University of New Mexico Cancer Center; Ducinea D Quintana, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- UNM Cancer Research and Treatment Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: UNM Cancer Center — http://cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Therapy: Pomalidomide: 1 tablet orally, daily for 21 days of a 28 day cycle (dose per cohort) Everolimus: 1 tablet orally for 21 days of a 28 day cycle (dose as per cohort) Dexamethasone 40 mg (20 mg >75yrs) orally, days 1, 8,15, 22 of a 28 day cycle
  Combination therapy: Following determination of the maximum tolerated dosages in the phase I portion of this study, all patients enrolled in the extension portion will receive the predetermined dosage combination of pomalidomide, everolimus and dexamethasone.
  Cycles will span 28 days. Dosage schedules will be:
  1. Everolimus daily for 28 days of a 28 day cycle;
  2. Pomalidomide daily for 21 days of a 28 day cycle
  3. Dexamethasone once weekly (on days 1,8,15,22) of a 28 day cycle.
Period: Overall Study
Arm/Group | Combination Therapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dosage (MTD)(Phase I)
Description: The Maximum Tolerated Dose (MTD) will be determined by first identifying the dose level at which >= 30% of patients experience a Dose Limiting Toxicity (DLT) according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, over a 28 day cycle. DLT will be defined based on the rate of drug-related grade 3-5, non-hematological adverse events experienced within the first 4 weeks (1 cycle) for each combined dosage scheme. The MTD will be defined as one dosage level below which DLT was observed in >= 30% of patients.
Time Frame: 2 years
Population: There was only one patient enrolled. The MTD could not be calculated based on one patient.
Arm/Group | Combination Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Toxicity Profile
Description: The toxicity profile will be described by specific adverse event rates among patients experiencing > grade 3 hematologic events (lasting >7 days) or grades 3-5 non-hematologic adverse events, according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, over a 28 day cycle. Specific events will be described as the numbers of patients experiencing them within each treatment cohort.
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Anti-tumor Effect
Description: Anti-tumor effect will be assessed based on serum protein electrophoresis (SPEP) of the monoclonal protein (M-protein) and plasma concentrations of K/L free light chains (FLC) after each 28-day cycle. Descriptive statistics will be used for this measurement.
  Complete response (CR): disappearance of any M-protein and FLC as measured by SPEP and/or FLC. Pre-existing plasmacytomas must have completely resolved.
  Partial response (PR): >50% reduction in M-protein and >50% reduction in the difference between involved and uninvolved FLC. Any plasmacytoma must have decreased in size by >50%.
  Stable disease: not meeting criteria for CR, PR, or progressive disease (PD). PD: >25% increase from baseline in serum or urine M-protein (serum M-protein must increase by > 0.5 gm/dl; urine M-protein must increase by >200 mg /24 hr); or development of new plasmacytomas or new lytic bone lesions; or a measurable increase in the size of these lesions; or hypercalcemia (>11.5 mg/dl) attributed to MM.
Time Frame: 3.5 years
Population: There was only one patient enrolled. Anti-tumor effect cannot be reported accurately based on results from one patient.
Arm/Group | Combination Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Response Rate (RR)
Description: ORR is the percentage of patients with a > Partial Response (PR). Response is assessed based on serum protein electrophoresis (SPEP) of the monoclonal protein (M-protein) and plasma concentrations of K/L free light chains (FLC) after each 28-day cycle.
  Complete response (CR): disappearance of any M-protein and FLC as measured by SPEP and/or FLC. Pre-existing plasmacytomas must have completely resolved.
  PR: >50% reduction in M-protein and >50% reduction in the difference between involved and uninvolved FLC. Any plasmacytoma must have decreased in size by >50%.
  Stable disease: not meeting criteria for CR, PR, or progressive disease (PD). PD: >25% increase from baseline in serum or urine M-protein (serum M-protein must increase by > 0.5 gm/dl; urine M-protein must increase by >200 mg /24 hr); or development of new plasmacytomas or new lytic bone lesions; or a measurable increase in the size of these lesions; or hypercalcemia (>11.5 mg/dl) attributed to MM.
Time Frame: 3 years
Population: There was only one patient enrolled. Response rates cannot be accurately reported based on one patient.
Arm/Group | Combination Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=1)
Alopecia (Hair loss) (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (hemoglobin levels decreased) (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 1 (6)
Headache (Nervous system disorders) | 1 (1)
Hypernatremia (high blood sodium) (Investigations) | 1 (1)
Hypoalbuminemia (low blood albumin) (Investigations) | 1 (1)
Hypokalemia (low blood potassium) (Investigations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Paresthesia (tingling, burning sensation) (Nervous system disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
White blood cell count decreased (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Low accrual led to early termination; only one subject was enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes